CLINICAL TRIAL: NCT06255535
Title: Repetitive Transcranial Magnetic Stimulation Guided by Personalized Brain Functional Sectors (pBFS) for Low-Functioning Autism Spectrum Disorder: a Multi-center, Randomized, Sham-controlled Trial
Brief Title: pBFS Guided rTMS Over Cognitive Control Network for ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changping Laboratory (Other)
Collaborators: Xi'an TCM Hospital of Encephalopathy (Unknown); Linyi Hedong Rehabilitation Hospital (Unknown); Jining Medical University (Other); Fujian Maternity and Child Health Hospital (Other); Fujian Children's Hospital (Unknown); Hebei Provincial Mental Health Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPASD05DL_Multicenter
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder
Keywords: intellectual or development delay; personalized; TMS; functional MRI
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active iTBS group (Experimental): active iTBS over DLPFC
  Interventions: Device: active iTBS treatment
- Sham group (Sham Comparator): sham iTBS over DLPFC
  Interventions: Device: sham iTBS treatment

INTERVENTIONS:
Device: active iTBS treatment — Participants will undergo three iTBS sessions per day, with 1800 pulses per session, over a 12-week period. Individualized targets will be generated using the pBFS technique.
  Arms: active iTBS group
Device: sham iTBS treatment — Participants will undergo three iTBS sessions per day, with 1800 pulses per session, over a 12-week period. Sham stimulation will be delivered through a sham coil with the identical appearance as real coil. Individualized targets will be generated using the pBFS technique.
  Arms: Sham group

SUMMARY:
The aim of this trial is to assess the efficacy and safety of precision neuromodulation for alleviating core symptoms in patients with autism spectrum disorder (ASD) who also have intellectual or developmental delay. The neuromodulation will be administered using intermittent theta burst stimulation (iTBS) targeting the left dorsolateral prefrontal cortex (DLPFC), guided by personalized Brain Functional Sector (pBFS) technology.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental condition characterized by impaired social communication and repetitive behaviors. Unfortunately, evidence-based treatments have not proven effective for older individuals with low-functioning ASD, despite their significant need for intensive support. However, emerging evidence suggests that Transcranial Magnetic Stimulation (TMS) has been successful in treating various psychiatric and neurological disorders.

Given the broad cognitive control dysfunction observed in ASD, targeting cognitive control function may offer a promising treatment approach. Leveraging the personalized Brain Functional Sector (pBFS) technique and task-free functional MRI scans, we can precisely locate the cognitive control function region within the left DLPFC, and follow-up at 24-week after initiation of treatment.

In this study, participants who meet the inclusion and exclusion criteria will be randomly assigned to either active or sham iTBS (intermittent theta burst stimulation) groups at a ratio of 2:1. The treatment protocol consists of a 12-week duration, with sessions conducted 5 days per week and 3 sessions iTBS over DLPFC per day. The inter-session interval is set at 30 minutes. Clinical evaluations focusing on ASD core symptoms and related behavioral profiles will be conducted at baseline and after the 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* 6-30 years old
* Have the diagnosis of autism spectrum disorder
* ADOS-2 score is higher than the ASD cut-offs
* Comorbid with intelligent disorder, IQ/DQ < 70
* Primary environmental language is Chinese
* Participant's parents or other legal guardians give informed consent

Exclusion Criteria:

* Genetic Disorders, such as (e.g., Down syndrome, Fragile X syndrome, Rett syndorme), Current or history of severe ADHD, tourette syndrome, psychotic disorders (e.g., schizophrenia, schizoaffective disorder, bipolar disorder)
* Severe self-injury or suicidal behavior exhibited within the past year
* Significant visual, auditory, deafness or motor disability that prevent them from following study procedures
* Current or history diagnosis of epilepsy
* Known severe physical diseases, particularly those affecting the brain
* Metal implantation contradicted by MRI or TMS, such as artificial cardiac pacemakers, stents, cochlear implants
* Respiratory or circulatory conditions increasing sedation risk, such as Apnea syndrome, severe snoring, or other relevant diseases
* All legal guardians are illiterate, unable to read informed documents or complete questionnaires independently
* Received transcranial magnetic stimulation (TMS), transcranial current stimulation (tCS), focused ultrasound (FUS), or other neuromodulation treatment in the last 3 months
* Current participation in other clinical trials

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 215 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
ADOS-2 SA CSS score change after treatment | Pre-treatment (baseline), post-treatment (12-week)
  The score changes of ADOS-2 SA CSS (Autism Diagnostic Observation Scale, 2nd edition, social affect domain, calibrated severity score) at 12-week from baseline. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
ADOS-2 SA CSS score change from baseline to follow-up | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  The score changes of ADOS-2 SA CSS from baseline, to 12-week posttreatment and, to 24-week follow-up. Higher scores mean a worse outcome.
Response rate in social ability after 12-week iTBS treatment | Pre-treatment (baseline), post-treatment (12-week)
  Treatment response is defined as improvement, i.e., at least 1-point decreased, in the ADOS-2 SA For ADOS-2 SA, higher scores means more severe symptom.
Response rate in social ability at 24-week follow-up | Pre-treatment (baseline), follow-up (24-week)
  Treatment response is defined as improvement, i.e., at least 1-point decreased, in the ADOS-2 SA For ADOS-2 SA, higher scores means more severe symptom.
ADOS-2 total CSS change with treatment | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  The ADOS-2 total CSS score change from baseline. Higher scores mean a worse outcome.
SCQ score change with treatment | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  The SCQ (Social Communication Questionnaire) score change from baseline. Higher scores mean a worse outcome.
CBCL score change with treatment | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  The CBCL (Child Behavior Checklist) score change from baseline. Higher scores mean a worse outcome.
QoL score change with treatment | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  The QoL (quality of life) score change from baseline. Higher scores mean a worse outcome.
AIM score change with treatment | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  The AIM (Autism Impact Measure) score change from baseline. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (6):
- China (6):
  - Fujian Children's Hospital, Fuzhou, Fujian
  - Fujian Maternity and Child Health Hospital, Fuzhou, Fujian
  - Hebei Provincial Mental Health Center, Baoding, Hebei
  - Xi'an TCM Hospital of Encephalopathy, Xi'an, Shaanxi
  - Jining Medical University, Jining, Shandong
  - Linyi Hedong Rehabilitation Hospital, Linyi, Shandong

IPD SHARING:
Plan to Share IPD: No